CLINICAL TRIAL: NCT06344403
Title: Clinical Efficacy and Safety of Tender Point Infiltration (TPI) for Management of Acute and Subacute Zoster Associated Pain
Brief Title: Clinical Efficacy and Safety of Tender Point Infiltration (TPI) for Acute and Subacute Zoster Associated Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Managrment, Beijing Tiantan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-045-02
Record Dates: First submitted 2024-03-17; First posted 2024-04-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Herpes Zoster; Local Infiltration; Acute Pain
Keywords: Herpes zoster; Acute pain
MeSH Terms: conditions — Herpes Zoster; Acute Pain | interventions — Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard gorup (Active Comparator): Patients will receive standard oral medicine for herpes zoster.
  Interventions: Drug: analgesic
- TPI group (Experimental): Patients will receive standard medicine treatment and tender point infiltrations therapy.
  Interventions: Drug: analgesic; Behavioral: Tender point infiltration

INTERVENTIONS:
Drug: analgesic — Patients will receive daily 300 mg pregabalin in divided doses (150 mg/12 hours). Once the patient report mild pain (VAS ≤ 3), the trial for reducing the pregabalin dose will be done. Nonsteroidal anti-inflammatory drug celecoxib (200 mg on request, up to two times daily)27 and tramadol (100 mg on request, up to 400mg daily) will be available for as-needed analgesia.
  Other Names: Standard treatment
Behavioral: Tender point infiltration — Lidocaine mixed with diprospan injected into tender points.
  Other Names: TPI infiltration
  Arms: TPI group

SUMMARY:
Herpes zoster (HZ) is a skin infection disease which cause severe zoster-associated pain (ZAP) along sensory nerve in the corresponding segment. Evidence for the efficacy of existing local therapies for acute/subacute ZAP is limited. The hypothesis is that patients with acute/subacute ZAP treated with TPIs with local anesthetic and steroids under the basis of standard treatment will show better clinical outcomes compared with subjects treated with standard antiviral medicine treatment only.

DETAILED DESCRIPTION:
The conventional therapies for HZ infection can be seen in two phases. Those in acute phase are mainly antiviral (acyclovir, famciclovir, etc.), analgesic drugs (opioids, acetaminophen or nonsteroidal anti-inflammatory agents, gabapentin, etc.), while these conventional drug therapies could yield potential side effects, and part of patients are not fully satisfied with the analgesic effect. It is considered that supplementary and alternative local therapies may have better results with less side effects and reduce medical costs to relieve pain associated with HZ infection. These options, including nerve blockade (epidural injection, paravertebral injection, sympathetic block, intercostal nerve block, intracutaneous injection), pulsed radiofrequency16, acupuncture, fire needling acupuncture, electrical nerve stimulation19, lidocaine patch, capsaicin cream, and botulinum toxin injection have been reported to give positive therapeutic effects on acute herpes zoster neuralgia (AHN), however, evidence for the efficacy of existing local therapies is limited and risks may occur due to high invasiveness of some procedures, there is insufficient evidence and expert agreement to make recommendations for these intervention strategies as first-line treatments in guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with onset of HZ rash less than 90 days.
2. HZ affected the spinal nerves (cervical/thoracic/lumbar nerve).
3. Aged 18 to 75 years (inclusive).
4. Pain intensity > 7 cm on a visual analogue scale (VAS 0-10 cm).
5. Agreed to sign the informed consent form.

Exclusion Criteria:

1. Infection at the puncture site.
2. Poor general situation unable to be treated.
3. A history of abuse of narcotics.
4. Non-compliance or inability to complete the self-evaluation questionnaires.
5. Pregnancy or lactation.
6. Patients using immunosuppressants and those with severe systemic diseases such as hematological malignancies, cancers, or autoimmune disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The presence of postherpetic neuralgia using VAS score | 12 months
  12 months after the treatments, number of patients with any pain with a VAS score of higher than 0/Number of all patients，0="no pain" and 10="worst pain imaginable"

SECONDARY OUTCOMES:
visual analogue scale score at each time point | before the treatment (baseline), 30min after the intervention (for TPI group), then 1 day, 2 weeks, 1 month, 3 months, 6 months and 12 months following the treatment
  0 = 'no pain at all' to 10 = 'worst pain imaginable'
Proportion of patients receiving repeated TPIs and block points | 12 months
  Number of patients receiving TPI treatments more than twice/Number of all patients
Consumption of oral drugs at each time point | day 1, then 2 weeks, 1 month, 3 months, 6 months and 12 months following the treatment.
  Dose of celecoxib, pregabalin and tramadol
The presence of PHN at month 3 and month 6 post treatment | 3 and 6 months after treatments
  Number of patients with any pain with a VAS score of higher than 0/Number of all patients (0 = 'no pain at all' to 10 = 'worst pain imaginable')
Patient satisfaction scores on the 5-point Likert scale | day 1, then week 2, month 1, month 3, month 6 and month 12 following the treatment
  1: Very dissatisfied,2: Dissatisfied,3: Not sure,4: Satisfied,5: Very satisfied
Quality of life on the Scores on the WHOQOL-BREF | day 1, then week 2, month 1, month 3, month 6 and month 12 following the treatment
  Scores on the WHOQOL-BREF. The responses are given on 5-point Likert scale (1-5) and the overall score ranges from 0 to 100; a higher score corresponds to better QoL.
Adverse reactions through study completion | After treatments
  Any side effect and uncomfortable situation related to treatment through study completion，an average of 1 year
Predictive factors for the prevention of PHN at month 12 posttreatment | month 12 posttreatment
  the correlation between patients' baseline characteristics and the incidence of PHN will be analyzed 12 months after treatment in TPI group.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.
Supporting Information: Study Protocol, CSR